CLINICAL TRIAL: NCT01933867
Title: Water-aided Colonoscopy in Patients With Inflammatory Bowel Disease - a Single-center, Single-blinded Randomized Trial
Brief Title: Water-aided Colonoscopy in Inflammatory Bowel Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitkovice Hospital (Other)
Responsible Party: Principal Investigator, Premysl Falt MD, MUDr. Premysl Falt, Ph.D., Vitkovice Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DDC VN 06
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-06

CONDITIONS: Inflammatory Bowel Disease
Keywords: water; colonoscopy; Crohn´s disease; ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water immersion colonoscopy (Experimental): Water immersion during colonoscope insertion and room air insufflation during colonoscope withdrawal.
  Interventions: Procedure: Water immersion
- Air insufflation colonoscopy (Active Comparator): Standard room air insufflation during both colonoscope insertion and withdrawal.
  Interventions: Procedure: Air insufflation insertion

INTERVENTIONS:
Procedure: Water immersion — Water immersion means infusion of room temperature water during colonoscope insertion without air insufflation.
  Arms: Water immersion colonoscopy
Procedure: Air insufflation insertion
  Other Names: Room air insufflation during colonoscope insertion.
  Arms: Air insufflation colonoscopy

SUMMARY:
Water-aided insertion of the colonoscope has been repeatedly proven to beneficial in terms of lower discomfort and need for sedation during colonoscopy. Patients with inflammatory bowel diseases (IBD) undergo repeated colonoscopy in course of their disease. According to our preliminary experience, water immersion could be beneficial while scoping these patients. As far as the investigators know, water-aided colonoscopy has never been studied in this indication. Results of our trial might support use of water-aided colonoscopy in common practice and decrease associated discomfort in IBD patients.

ELIGIBILITY:
Inclusion Criteria:

* known diagnosis of inflammatory bowel disease
* planned diagnostic outpatient colonoscopy
* signed informed consent
* willingness to undergo unsedated colonoscopy

Exclusion Criteria:

* ulcerative proctitis
* bowel resection longer than ileocecal resection
* requirement for sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Success rate of unsedated colonoscopy | at the end of each colonoscopy
  Successful unsedated colonoscopy is defined as reaching the cecum by using given insertion technique without administering sedation.

SECONDARY OUTCOMES:
Discomfort during colonoscopy | at the end of each colonoscopy
  Discomfort level using visual continuous scale 0-10 (0 = no pain, 10 = worst pain).
Cecal intubation time | while reaching the cecum
  Cecal intubation time is defined as time between colonoscope introduction into the anus and reaching the cecum.

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Diseases Center, Vitkovice Hospital, Ostrava, Czechia

REFERENCES:
- [Derived] Falt P, Smajstrla V, Fojtik P, Urban O, Hill M. Water-Aided Colonoscopy in Inflammatory Bowel Disease Patients-A Randomised, Single-Centre Trial. J Crohns Colitis. 2015 Sep;9(9):720-4. doi: 10.1093/ecco-jcc/jjv093. Epub 2015 Jun 3. PMID 26040317